

جامىعة محمدين راشىد للطب والعلوم الصحية Mohammed Bin Rashid University of Medicine and Health Sciences

## Institutional Review Board (MBRU-IRB) Patient Information Sheet/Informed Consent

## Informed Consent to Participate in a Research Study 25 August 2024

1. Study Title: Accuracy of intraorally scanned denture impressions compared to conventional border molded impressions- in vivo study

The above-mentioned study has been approved by the Dubai Scientific Research Ethics Committee, DHA]

**Principal Investigator:** Dr. Fatemeh Amir Rad

Address: Hamdan Bin Mohammad College of Dental Medicine (HBMCDM) at Mohammad Bin Rashid

University of Medicine and Health Sciences (MBRU).

Building No 34, Dubai Health Care City

Dubai - UAE

Phone: +971 4 383 8910

Site where the study will be conducted: Dubai Dental Hospital

You are invited to participate in this research study conducted at Hamdan Bin Mohammad College of Dental Medicine/ Dubai Dental Hospital - Dubai Health. Please, take your time to read the following information carefully, before you decide whether you wish to take part in this research study or not. You are encouraged to ask the study investigator if you need any additional information or clarification about what is stated in this form and/or in the research study as a whole. You are also free to take this information sheet and consult with your doctor or other health professionals. Please note that, should you decide to participate, you are free to withdraw at any time without any consequence.

### The purpose of the Research Study and Overview of Participation

The purpose of this study is to evaluate the accuracy of an intra oral scanner digital impression in a completely edentulous arch and compare it with a conventional impression.

All patients attending Dubai Dental Hospital for complete denture treatment will be invited to participate in this study.

| Form Number | Version | Referenced Policy | Last Review | Page No. |
|-------------|---------|-------------------|-------------|----------|
| RGS F010 | 3.0 | RGS-P001 | May-2023 | 1 of 4 |



جامىعة محمدين راشيد للطب والعلوم الصحية Mohammed Bin Rashid University of Medicine and Health Sciences

## Institutional Review Board (MBRU-IRB) Patient Information Sheet/Informed Consent

#### What is the duration of the study?

Around two months

### Participation in the study – Why participate, what will happen on participation, what is required of the patient.

Participation in this study will provide the investigators with scientific data to validate alternative digital impression obtaining methods.

The process of denture provision will be the same, however, at the impression taking stage, two methods of impression capturing will be performed.

#### Any Risks as a Result of Participating in the Study

There are no risks associated with participation in the study except for longer chair time which wi communicated to them prior to consenting to participation. Participants will have the right to stop impression capturing procedure or withdraw from the research at any time.

#### Any Benefits as a Result of Participating in the Study

The data collection is part of the process of complete denture provision to the patients.

#### **Any Alternative Treatment**

N/A

If you agree to take part in this research study, please, be assured that the obtained information will be kept confidential. Unless required by law, only the study investigator or designee, the MBRU-Institutional Review Board (MBRU-IRB), the Dubai Scientific Research and Ethics Committee (DSREC) and/or inspectors from governmental agencies will have direct access to your information.

'If you are harmed by taking part in this research project, there are no special compensation arrangements. If you are harmed due to someone's negligence, or have any concerns about any aspect of the way you have been approached or treated during the course of this study, you can contact Dubai Scientific Research Ethics Committee, DHA on 800 342 or email on DSREC@dha.gov.ae

| Form Number | Version | Referenced Policy | Last Review | Page No. |
|-------------|---------|-------------------|-------------|----------|
| RGS F010 | 3.0 | RGS-P001 | May-2023 | 2 of 4 |



جام<u>عة محمدين راشح</u> للطب والعلوم الصحية Mohammed Bin Rashid University of Medicine and Health Sciences

### **Institutional Review Board (MBRU-IRB) Patient Information Sheet/Informed Consent**

3 of 4

May-2023

RGS F010

3.0

| Investigator's Statem | ent: | | | | |
|---|---|---|---|---|---|
| | al representati<br>ered all the pa | ve, or parent/guard | ian) the pu | irpose of the | dy with<br>study and its risks and<br>e participant in case of |
| Name of Investigator | or Designee | Signature | C | Date & Time | |
| Patient's Participation | <u>n:</u> | | | | |
| I voluntarily agree to Rad at 04 383 8910 or If I feel that my ques understand that secti Dubai Dental Hospita I give permission for withdraw this consentorm, and it will not a consent. | be a part of the any of his/her tions have not ons of any of n l or from regulathese individuct and disconting ffect my care of | is research study are team involved in the been answered, I do not make the been at the been at the bear at the bear the benefits. I know the benefits. I know the benefits. I know the benefits. | an contact an contact by be looke are it is re to my reco this projec | hat I can cont<br>case I have and<br>the DSREC (I<br>d at by respond<br>levant to my t<br>rds. I unders<br>t at any time, | s have been answered. act Dr. Fatemeh Amir ny questions. OSREC@dha.gov.ae). I nsible individuals from aking part in research. tand that I am free to even after signing this of this signed informed |
| I agree to take part in | the above stu | dy. | | | |
| Name of Patient/Legal<br>Representative or<br>Parent/Guardian | | Signature | | Date & Time | |
| Form Number | Version | Referenced Pol | cy | Last Review | Page No. |

RGS-P001



جام<u>عة محمدين راشح</u> للطب والعلوم الصحية Mohammed Bin Rashid University of Medicine and Health Sciences

# Institutional Review Board (MBRU-IRB) Patient Information Sheet/Informed Consent

| Name of the Witness<br>(if patient, representative<br>or parent does not read) | Witness's Signature | Date & Time |
|---|---|---|

| Form Number | Version | Referenced Policy | Last Review | Page No. |
|-------------|---------|-------------------|-------------|----------|
| RGS F010 | 3.0 | RGS-P001 | May-2023 | 4 of 4 |